CLINICAL TRIAL: NCT05231291
Title: Association Between Handgrip Strength, Skinfold Thickness and Trunk Strength Among University Students
Brief Title: Association Between Handgrip Strength, Skinfold Thickness and Trunk Strength
Status: Completed | Type: Observational
Sponsor: King Khalid University (Other)
Responsible Party: Principal Investigator, Snehil Dixit, Assistant Professor, King Khalid University
Other Study IDs: ECM#2021-3603
Record Dates: First submitted 2022-01-19; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Young Adult
Keywords: Hand Grip Strength; Skinfold Thickness; Trunk strength
MeSH Terms: interventions — Hand Strength

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young Adults: Skinfold thickness (SFT) at multiple marked sites on biceps, triceps, subscapular and suprailiac areas using a Harpenden Caliper (Baty, UK) for the non-dominant side.
  Hand grip strength measurement Jamar Hydraulic Dynamometers (Hydraulic Hand Dynamometer Fabrication Enterprises Inc, NY) was used as the evaluation tool for measuring grip.
  The handgrip measurement was carried out as per the recommendations laid by The National Institute of Health Research (NIHR).
  The T score for hand grip strength was also calculated. Also the mean predicted handgrip strength for given height was calculated foe the given height Trunk muscle strength testing was done. An analogue hydraulic push-pull dynamometer (Model: FEI-12-0394) was used to evaluate. The trunk extensor and flexor muscle strength was evaluated using and was recorded in pounds (lbs.).
  Interventions: Other: hand grip strength

INTERVENTIONS:
Other: hand grip strength — Observational study
  Other Names: trunk strength; skinfold measurement

SUMMARY:
The main objective was to explore relationship between skinfold measurement at multiple sites, hand grip strength, and trunk muscle strength (flexors and extensors) in healthy participants. Conclusion: There is a moderate association between hand grip strength, T score and trunk muscle strength, evident from the present research. Though no such association was seen for skinfold measurement.

DETAILED DESCRIPTION:
Objectives: The main objective was to explore relationship between skinfold measurement at multiple sites, hand grip strength, and trunk muscle strength (flexors and extensors) in healthy participants. Methods: Cross-sectional design, randomly recruited 40 participants. Finally only 39 participants were included. Measurements for demographic variable and anthropometric variables were done. Then the evaluation for hand grip strength and skin fold was done. Data Analysis: Quantitative variables were designated using means and standard deviations, and qualitative variables described by frequencies. The Repeated measure for Analysis of Variance (RANOVA) was used to analyse whether there was statistically significant interaction between the two groups (smoking vs non-smokers). The Pearson correlation coefficient was used to measure associations of anthropometric traits with grip strength. Multiple linear regression model was also carried to explore the linear relationship between dependent and independent variables.

ELIGIBILITY:
Inclusion Criteria:

* This cross-sectional study Only healthy participants with no known history of previous diseases were included (n=39).

Exclusion Criteria:

* Students who found it difficult to follow the instructions for the tests after one familiarity sessions were excluded (n=0). Students reporting any kind of acute infections, previous history of chronic respiratory diseases were also excluded (n=1).

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Young Adults Age between 18-25 Graduate students
Study Population: College students within the age group of 18-25 years. We were interested in looking for Association between hand grip strength , Skinfold thickness and trunk strength
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Handgrip strength | 1 month
  Jamar Hydraulic Dynamometers (Hydraulic Hand Dynamometer Fabrication Enterprises Inc, NY) was used as the evaluation tool for measuring grip.
  The handgrip measurement was carried out as per the recommendations laid by The National Institute of Health Research (NIHR)
Trunk strength | 1 month
  Hydraulic Dynamometers (Hydraulic Dynamometer)
Skinfold thickness | 1 month
  Harpenden Caliper , Skinfold thickness (SFT) at multiple marked sites on biceps, triceps, subscapular and suprailiac areas using a Harpenden Caliper (Baty, UK) for the non-dominant side. The instruments were well calibrated before testing. The measurement sites were marked, and then a minimum of two readings were taken. In case the two measurements at a particular site differed by more than 3 mm, a third measurement was taken. The mean of the two closest measurement was documented and the percentage of body fat was then calculated using the formula and table published by Durnin and Womersley

SECONDARY OUTCOMES:
Waist Circumference | 1 month
  Waist circumference was measured using inch tape as per the guidelines laid by the world health organization (WHO) . Elements of the protocol discussed below include:
  * the anatomical placement of the measuring tape, its tightness and the type of tape used;
  * the subject's posture, phase of respiration, abdominal tension, stomach contents and clothing.
Smoking Habits | 1 month
  Yes and No type questions , have been chronic smokers of more than 1 year or 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- King Khalid University, Abhā, 'Asir Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
As per the Regulation from King Khalid University